CLINICAL TRIAL: NCT03524716
Title: Self-monitoring and Reminder Texts to Increase Physical Activity After Cancer II (Smart Pace II)
Brief Title: Self-monitoring and Reminder Texts to Increase Physical Activity After Cancer II
Acronym: SmartPaceII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 174525; NCI-2018-00621 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-04-04; First posted 2018-05-15 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: physical activity; digital health; text messages; intervention; exercise; randomized; Fitbit
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit and Text Messages (Experimental): Participants randomized to this arm receive print materials and a Fitbit Flex 2 at baseline and daily text messages for 12 weeks.
  Interventions: Behavioral: Fitbit and Text Messages
- Usual Care (No Intervention): Participants randomized to usual care receive print materials at baseline.

INTERVENTIONS:
Behavioral: Fitbit and Text Messages — Physical activity tracker wristband and daily text messages delivered to the participants' phones.
  Arms: Fitbit and Text Messages

SUMMARY:
There is a critical need for physical activity interventions in colorectal cancer (CRC). The investigators have developed a digital health physical activity intervention, Smart Pace, which includes a wearable tracker (Fitbit) and text messaging and aims to have patients build up to 150 min/wk of moderate activity. In this study, the investigators propose to expand and improve Smart Pace, including: 1) enrolling patients during chemotherapy; 2) tailoring text messages to individual preferences and treatment timing; and 3) adding resources to support home-based exercise. The study is a 12-week pilot randomized controlled trial (RCT) to evaluate the feasibility of this novel digital health physical activity intervention among 48 CRC patients on chemotherapy. The specific aims are to: 1) Determine the feasibility of the intervention via adherence and attrition, and determine the acceptability of the intervention via questionnaires and semi-structured interviews . 2) Estimate the effect of the intervention vs. usual care on physical activity, QOL, and symptoms at 12-weeks . And 3) Explore the impact of the intervention vs. usual care on fitness, weight, waist circumference, and blood pressure at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colon or rectal adenocarcinoma
* Expected to receive at least 12 weeks of chemotherapy
* Able to speak and read English
* Access to a mobile phone with Internet and text messaging capabilities
* ≥4 weeks since last major surgery and fully recovered
* ≥18 years old
* Physician consent to participate in unsupervised moderate intensity physical activity
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Engaging in 150 minutes/week or more of moderate physical activity, 75 minutes/week or more of vigorous physical activity, or an equivalent combination
* Hypertension that is not well-controlled (≥160/90) on anti-hypertensive therapy
* Any contraindications to exercise, including, but not limited to: brain metastases; current congestive heart failure (New York Heart Association Class II, III or IV); serious or nonhealing wound, ulcer, or bone fracture; spinal cord compromise or instrumentation due to metastatic disease; peripheral neuropathy ≥grade 3; advanced Chronic Obstructive Pulmonary Disease (COPD) on oxygen
* Serious cardiovascular event within 6 months including, but not limited to, transient ischemic attack (TIA), cerebrovascular accident (CVA), or myocardial infarction (MI)
* Has been told by a doctor that he/she has a heart condition and recommended to only engage in medically supervised activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Fitbit wear time | up to 12 weeks from study start
  Number of study days Fitbit is worn
Acceptability of the intervention | At 12 weeks from study start
  Acceptability will be assessed with an investigator created questionnaire among participants in the intervention arm.
Text message response rate | up to 12 weeks from study start

SECONDARY OUTCOMES:
Objective physical activity | At 0 weeks and 12 weeks from study start
  Minutes of moderate-to-vigorous physical activity per week measured by accelerometer
Fatigue | At 0 and 12 weeks from study start
  Lee Fatigue Scale
Cardiorespiratory fitness | At 0 and 12 weeks from study start
  6 minute walk test
Anthropometrics, Waist circumference | At 0 and 12 weeks from study start
Anthropometrics, Body weight | At 0 and 12 weeks from study start
Sleep quality | At 0 and 12 weeks from study start
  Will be assessed by the Pittsburgh Sleep Quality Index, providing a score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Health-related quality of life in cancer patients | At 0 and 12 weeks from study start
  Will be assessed via the European Organization for Research and Treatment (EORTC) of Cancer Quality of Life Questionnaire-Core 30
Health-related quality of life in colorectal cancer patients | At 0 and 12 weeks from study start
  Will be assessed via the European Organization for Research and Treatment (EORTC) of Cancer Quality of Life Questionnaire-Core 29
Neuropathy | At 0 and 12 weeks from study start
  Will be assessed by the Chemotherapy-Induced Peripheral Neuropathy 20 (CIPN20) questionnaire, a 20-item quality of life questionnaire.
Anxiety | At 0 and 12 weeks from study start
  Will be assessed by the Spielberger State-Trait Anxiety Inventories (STAI), consisting of 40 questions on a self-report basis. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Depression | At 0 and 12 weeks from study start
  Will be assessed by the Center for Epidemiological Studies-Depression Scale (CES-D), a brief self-report questionnaire which consists of 20 questions. Scores on the CES-D range from 0 to 60, in which higher scores suggest a greater presence of depressive symptoms.
Leisure-time physical activity | At 0 and 12 weeks from study start
  Will be assessed via the Harvard Health Professionals Follow-up Study (HPFS) physical activity questionnaire.
Perceived barriers to physical activity | At 0 and 12 weeks from study start
  Modified from the Project Graduate Ready for Activity Daily(GRAD) survey - 24 items plus a write-in option.
Exercise Confidence | At 0 and 12 weeks from study start
  Modified from the Project GRAD (Graduate Ready for Activity Daily) survey - 11 items.
Social support | At 0 and 12 weeks from study start
  Modified from the Project GRAD (Graduate Ready for Activity Daily) survey - 13 items asked about social support.

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Van Blarigan, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Results from this pilot clinical trial will be reported at national conferences and published in peer-review journals.

REFERENCES:
- [Derived] Van Blarigan EL, Dhruva A, Atreya CE, Kenfield SA, Chan JM, Milloy A, Kim I, Steiding P, Laffan A, Zhang L, Piawah S, Fukuoka Y, Miaskowski C, Hecht FM, Kim MO, Venook AP, Van Loon K. Feasibility and Acceptability of a Physical Activity Tracker and Text Messages to Promote Physical Activity During Chemotherapy for Colorectal Cancer: Pilot Randomized Controlled Trial (Smart Pace II). JMIR Cancer. 2022 Jan 11;8(1):e31576. doi: 10.2196/31576. PMID 35014958